

# Patient Adherence to Lung Cancer Screening Patient Interview

| Principal Investigator: Robert | J. Volk, PhD |
|--------------------------------|--------------|
| Participant's Name | Study ID |

# **Study Purpose**

The goal of this behavioral research study is to understand participants' barriers to lung cancer screening and their experience with scheduling lung cancer screening.

You are being asked to take part in this study because you may be eligible for lung cancer screening at the UTMB Comprehensive Lung Cancer Screening Program and the UT Health East Texas Lung Nodule Program.

# **Study Procedures**

If you agree to take part in this study, you will participate in an interview. During the interview, you may be asked about:

- Your background information, such as your race and level of education
- Your lung cancer diagnosis and your history of lung cancer screening
- Your experience with scheduling lung cancer screening
- Any barriers that kept you from completing screening
- Ideas that might make screening completion easier

#### Length of the Study

Your participation will be over after you complete the interview, which may take up to 1 hour.

#### **Potential Risks**

Surveys may contain questions that are sensitive in nature. You may feel uncomfortable when answering some of the survey questions. You may refuse to answer any questions that make you feel uncomfortable.

The research team does not expect you to experience any significant risks in participating in this study, but this study may involve unpredictable risks to the participants. If you have concerns about completing the surveys, you are encouraged to contact your doctor or the study chair.

#### **Potential Benefits**

There are no benefits to you from your taking part in this research. Future patients may benefit from what is learned.

## **Costs and Compensation**

There will be no cost to you for taking part in this study. As compensation for your time



and effort, you will be mailed a \$100 gift card after you complete the surveys.

# **Voluntary Participation**

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

# Confidentiality

To maintain confidentiality, any information that could be used to identify you will be stored securely online or in locked files. Any information that could identify you will be removed or changed before results are made public.

### **Future Research**

After personal information is removed, your information could be distributed to another investigator or used for future research studies without additional informed consent.

There is a possibility that you might be contacted in the future about this study or other research opportunities, but that you may refuse any further participation if you wish.

# **Number of Participants**

Up to 30 patients from the UTMB Comprehensive Lung Cancer Screening Program and the UT Health East Texas Lung Nodule Program will take part in this study.

# **Funding**

This research is funded by the Cancer Prevention and Research Institute of Texas.

#### **Questions or Concerns**

If you have questions, concerns, or think the research has hurt you, talk to the research team at 713-563-0020. If you want contact someone independent of the research team, contact the Institutional Review Board at (713) 792-6477.

# **Sharing of Protected Health Information**

During the course of this study, the research team at The University of Texas MD Anderson Cancer Center will be collecting information about you that they may share with health authorities, study monitors who check the accuracy of the information, and individuals who put all the study information together in report form. By agreeing to take part in this study, you are providing authorization for the research team to use and share your information at any time. If you do not want to authorize the use and disclosure of your information, you may choose not to take part in this study. There is no expiration date for use of this information. You may withdraw your authorization at any time, in writing, for any reason as long as that information can be connected to you. You can learn more about how to withdraw your authorization by calling the Chief Privacy Officer at 713-745-6636 or by contacting the principal investigator at 713-563-0020 with any questions you have about the study.

## **Document Consent**

Before you can take part in this study, you must agree to the following statement:



I have been given the description of the study, my questions (if any) have been answered to my satisfaction, and I have decided to take part in the research study described here. [Circle one]

Yes No



# Patient Adherence to Lung Cancer Screening Patient Survey

| Principal Investigator: Robert J. Vo | lk, PhD |
|--------------------------------------|----------|
| Participant's Name | Study ID |

# **Study Purpose**

The goal of this behavioral research study is to understand participants' barriers to lung cancer screening and their experience with scheduling lung cancer screening.

You are being asked to take part in this study because you are eligible for lung cancer screening at the UTMB Comprehensive Lung Cancer Screening Program or the UT Health East Texas Lung Nodule Program.

# **Study Procedures**

If you agree to take part in this study, you will participate in answering a 5-part survey. You will be able to fill out this survey online or on paper (by mail). During the surveys, you may be asked about:

- Your background information, such as your race and level of education
- Lung cancer and your history of lung cancer screening
- Questions about screening reminders or navigation you may have received at your program

#### Length of the Study

Your participation will be over after you complete the surveys, which may take up to 1 hour.

#### **Potential Risks**

Surveys may contain questions that are sensitive in nature. You may feel uncomfortable when answering some of the survey questions. You may refuse to answer any questions that make you feel uncomfortable.

The research team does not expect you to experience any significant risks in participating in this study, but this study may involve unpredictable risks to the participants. If you have concerns about completing the surveys, you are encouraged to contact your doctor or the study chair.

#### **Potential Benefits**

There are no benefits to you from your taking part in this research. Future patients may benefit from what is learned.

## **Costs and Compensation**



There will be no cost to you for taking part in this study. As compensation for your time and effort, you will be mailed a \$25 gift card after you complete the surveys.

# **Voluntary Participation**

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

There is a possibility that you might be contacted in the future about this study or other research opportunities, but that you may refuse any further participation if you wish.

# Confidentiality

Any information that could be used to identify you will be stored securely online or in locked files. Any information that could identify you will be removed or changed before results are made public.

#### **Future Research**

After personal information is removed, your information could be distributed to another investigator or used for future research studies without additional informed consent.

# **Number of Participants**

Up to 300 patients from the UTMB Comprehensive Lung Cancer Screening Program and up to 300 patients from the UT Health East Texas Lung Nodule Program will take part in this study.

## **Funding**

This research is funded by the Cancer Prevention and Research Institute of Texas.

#### **Questions or Concerns**

If you have questions, concerns, or think the research has hurt you, talk to Dr. Robert J. Volk and the research team at 713-563-0020. If you want contact someone independent of the research team, contact the Institutional Review Board at (713) 792-6477.

# **Sharing of Protected Health Information**

During the course of this study, the research team at The University of Texas MD Anderson Cancer Center will be collecting information about you that they may share with health authorities, study monitors who check the accuracy of the information, and individuals who put all the study information together in report form. By agreeing to take part in this study, you are providing authorization for the research team to use and share your information at any time. If you do not want to authorize the use and disclosure of your information, you may choose not to take part in this study. There is no expiration date for use of this information. You may withdraw your authorization at any time, in writing, for any reason as long as that information can be connected to you. You can learn more about how to withdraw your authorization by calling the Chief Privacy Officer at 713-745-6636 or by contacting the principal investigator at 713-563-0020 with any questions you have about the study.



# **Document Consent**

Before you can take part in this study, you must agree to the following statement:

I have been given the description of the study, my questions (if any) have been answered to my satisfaction, and I have decided to take part in the research study described here. [Circle one]

Yes No



# Patient Adherence to Lung Cancer Screening Lung Cancer Screening Program Directors and Staff Interviews

Principal Investigator: Robert J. Volk, PhD

# **Study Purpose**

The goal of this behavioral research study is to understand the facilitators of and barriers to achieving higher lung cancer screening adherence rates. This will be done through interviewing program directors and staff from UTMB Comprehensive Lung Cancer Screening Program (CLSP) in the Department of Pulmonary Critical Care & Sleep Medicine and the UT Health East Texas (UT Tyler) Lung Nodule Program.

#### **Study Procedures**

If you agree to take part in this study, you will complete a survey and participate in an interview. During the survey and interview, you may be asked about:

- Your role and length of employment at your institution
- Lung cancer and lung cancer screening
- Facilitators and barriers to lung cancer screening adherence at your program
- Your opinion on your institution's readiness to implement change

# Length of the Study

Your participation will be over after you complete the survey and interview, which may take up to 1 hour in total.

#### **Potential Risks**

Surveys may contain questions that are sensitive in nature. You may feel uncomfortable when answering some of the survey questions. You may refuse to answer any questions that make you feel uncomfortable.

The research team does not expect you to experience any significant risks in participating in this study, but this study may involve unpredictable risks to the participants. If you have concerns about completing the surveys, you are encouraged to contact your doctor or the study chair.

As an MD Anderson employee, your participation or non-participation in this study will not affect your employment status at the institution or your employee benefits. You will not be impacted (favorably or unfavorably) based on your study participation decision. None of the following will be affected:

- Performance evaluations
- Career advancement
- Assignments
- Time off approvals

### **Potential Benefits**

There are no benefits to you from your taking part in this research. Future patients may



benefit from what is learned.

# **Costs and Compensation**

There will be no cost to you for taking part in this study. You will not receive any compensation for taking part in this study.

# **Voluntary Participation**

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

# Confidentiality

Any information that could be used to identify you will be stored securely online or in locked files. Any information that could identify you will be removed or changed before results are made public.

#### **Future Research**

After personal information is removed, your information could be distributed to another investigator or used for future research studies without additional informed consent.

There is a possibility that you might be contacted in the future about this study or other research opportunities, but that you may refuse any further participation if you wish.

# **Number of Participants**

Up to 10 directors and/or staff from the UTMB Comprehensive Lung Cancer Screening Program and the UT Health East Texas Lung Nodule Program will take part in this study.

# Funding

This research is funded by the Cancer Prevention and Research Institute of Texas.

#### **Questions or Concerns**

If you have questions, concerns, or think the research has hurt you, talk to the research team at 713-563-0020. If you want contact someone independent of the research team, contact the Institutional Review Board at (713) 792-6477.

#### **Document Consent**

Before you can take part in this study, you must agree to the following statement:

I have been given the description of the study, my questions (if any) have been answered to my satisfaction, and I have decided to take part in the research study described here. [Circle one]

Yes

No